CLINICAL TRIAL: NCT05423990
Title: Electroclinical Features of Sudden Unexpected Death in Epilepsy (SUDEP) : a Multi-center Observational Study
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Liu Yonghong (Other)
Responsible Party: Sponsor-Investigator, Liu Yonghong, professor, Xijing Hospital
Organization: Xijing Hospital (Other)
Other Study IDs: KY20222037-C-1
Record Dates: First submitted 2022-06-14; First posted 2022-06-21 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Sudden Unexpected Death in Epilepsy; Near-Sudden Unexpected Death in Epilepsy
MeSH Terms: conditions — Sudden Unexpected Death in Epilepsy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Video-Electroencephalography — Three types of video EEG monitoring equipment produced by Nicolet, Bio-logic and Nihon Kohden were used to collect data in the multi-center. The 19-lead recording electrode was placed according to the international 10-20 system, and the average lead was used. The recording time was 24h. All patients underwent eyes open and closed test, intermittent photic stimulation and hyperventilation induction test.

SUMMARY:
Sudden unexpected death in epilepsy (SUDEP) is regarded as a leading cause of premature death in epilepsy patients. We aim to capture the whole process of SUDEP and near-SUDEP occurrence in patients with epilepsy, and expolre video-electroencephalograph (V-EEG) changes and marker. A Chinese multicenter study was carried out to determine electroencephalo-graph marker related to SUDEP to provide a scientific basis for the prevention of SUDEP in patients with epilepsy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with epilepsy who meet SUDEP or near-SUDEP diagnosis,
* Giving written informed consent to participate in the study from relatives or caregivers.

Exclusion Criteria:

* Refusing to recruitment from relatives or caregivers.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with epilepsy who experience SUDEP or near-SUDEP identified in a multicenter study between April 2022 and April 2024.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
The occurrence of SUDEP or near-SUDEP | 2022.04.01-2024.04.01
  Baseline, clinical characteristics and EEG markers of SUDEP patients were collected.

CONTACTS AND LOCATIONS:
Locations (1):
- Liu Yonghong, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Undecided